CLINICAL TRIAL: NCT06785311
Title: Native Spirit: Culturally-grounded Substance Use Prevention for Indigenous Adolescents
Brief Title: Native Spirit: Significant Aim 3: Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Amanda Hunter, Assistant Professor, Arizona State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020073
Record Dates: First submitted 2025-01-11; First posted 2025-01-21 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Substance Use; Self Esteem; Youth Drinking; Prevention, Suicide
Keywords: American Indian; Adolescent Health; Prevention; After-School Programs
MeSH Terms: conditions — Substance-Related Disorders; Underage Drinking; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Wait-list controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive the intervention (Native Spirit after-school program). Each intervention session is based on an Indigenous cultural value and cultural activity/practice that is specific to the community. The intervention is 10, 1.5 hour sessions that occur once/week from January-May 2025.
  After the Crossover the Intervention group will engage in "usual programming" August-December 2025.
  Interventions: Behavioral: Native Spirit After-School Program
- Wait-List Group (Active Comparator): The wait-list group will receive control or "usual" programming. Usual programming includes a life skills program that focuses on financial wellness for teens, called "Money Matters" (Usual Practice). Participants will learn valuable financial life skills. Control sessions will be facilitated by the research site partner (after-school program employees) who typically implement their usual programming. Control sessions will be held at the research site. Each control session will last for 60-90 minutes, once a week for 10 weeks taking place from August 2025 - December 2025
  After the Crossover the wait-list group will receive the intervention January-May 2026.
  Interventions: Behavioral: Native Spirit After-School Program

INTERVENTIONS:
Behavioral: Native Spirit After-School Program — Native Spirit is a culturally-grounded after-school program that is community-specific. The program is 10-sessions/weeks long and each session is 1.5-2 hours in duration. Each session is guided by a local cultural knowledge holder and is focused on a different cultural value and accompanying cultural practice. Native Spirit aims to promote self-esteem, cultural efficacy, awareness of cultural connectedness, and resilience while preventing and/or slow down the initiation of substance use.
  Other Names: Native Spirit

SUMMARY:
The proposed research will used community-based participatory research methods in an urban-based American Indian (AI) community to adapt, implement, and evaluate an after-school program, called Native Spirit (NS), that seeks to improve cultural identity, self-esteem, resilience, and prevent substance use by increasing cultural engagement. Prior research suggests that AI youth that are culturally engaged experience better health outcomes. Additionally, the use of culturally-specific after-school programs has been shown to increase feasibility and sustainability of prevention programs. In order to achieve the goals of this proposed study, the Principal Investigator (PI) will work with local community members and existing tribal partners to implement the 10-session culturally-grounded after-school program and evaluate the program with the following aims:

Specific Aim 3 (R00): Examine the effectiveness of NS (increases exposure to local cultural values and activities), a program that seeks to prevent or decrease substance use by strengthening self-esteem, resilience, and cultural identity with 2 Indigenous communities in Arizona using a wait-list control design with 3 data collection timepoints and participant interviews.

DETAILED DESCRIPTION:
Specific Aim (SA) 3:

The objective of SA 3 is to examine the effectiveness of Native Spirit (NS) in the Salt River Pima Maricopa Indian Community (SRPMIC) and Pascua Yaqui Tribe (PYT) adolescents (grades 7-12) on preventing or decreasing substance use and strengthening cultural identity, self-esteem, and resilience. SA 3 will use a wait-list control design.

Procedure:

Step 1: Recruitment and Consent 1.1 Recruitment and consent process will occur December 2024-January 2025 for SRPMIC and May-July2025 for PYT.

Step 2: Baseline Assessment - Time 1 (T1)

2.1 SRPMIC participants will take the T1 assessment in January 2025. Surveys will be conducted virtually on participant cell phones. The research team will also print out multiple hard copies of the survey for participants who do not have access to a cell phone. Participants will sit at individual desks that are spaced so they cannot see each others assessment answers to minimize confidentiality risks. PYT participants will take the T1 assessment in August 2025.

Who: Virtual surveys will be administered by the PI and research team. Where: T1 assessment will be completed at the research sites - the SRPMIC Way of Life Facility and the PYT Boys & Girls Club.

How Long: T1 assessment will take 20-30 minutes to complete. How/What data: T1 assessment data will be collected virtually through REDCap. Duration: T1 assessment data will be completed in January 2025 for SRPMIC and August 2025 for PYT.

Step 3: Spring 2025 Intervention 3.1 SA3 uses a wait-list control design. The SRPMIC will be allocated to the intervention first. This is because the PI has worked with the SRPMIC for five years and the SRPMIC already has a developed intervention curriculum (the PI will submit a modification for review once curriculum is updated for 2025 intervention). This will allow the PI and the PYT to adapt the intervention. The intervention group (SRPMIC) will receive the intervention (NS program). Each intervention session is based on an Indigenous cultural value and cultural activity/practice that is specific to the SRPMIC.

Who: Intervention sessions will be facilitated by local cultural knowledge holders. At least one member of the research team will attend each session to ensure fidelity Where: Intervention sessions will be held at the research sites - the SRPMIC Way of Life Facility How Long: Each intervention session will last for 60-90 minutes, once a week for 10 weeks Duration: The Spring intervention will take place from January 2025 - May 2025

3.2 The research team will take candid pictures during the intervention that can be used for results dissemination. Any identifiable pictures with youth who do not have signed assent/consent forms will be immediately deleted.

Step 4: Follow-Up Assessment - Time 2 (T2) 4.1 SRPMIC participants will take the T2 assessment in May 2025. Surveys will be conducted virtually on participant cell phones. The research team will also print out multiple hard copies of the survey for participants who do not have access to a cell phone. Participants will sit at individual desks that are spaced so they cannot see each other's assessment answers to minimize confidentiality risks.

Who: Virtual surveys will be administered by the PI and research team. Where: T2 assessment will be completed at the research site - the SRPMIC Way of Life Facility How Long: T2 assessment will take 20-30 minutes to complete. How/What data: T2 assessment data will be collected virtually through REDCap. Duration: The T2 assessment will be completed in May 2025

Step 5: Spring Participant interviews

5.1 Participants who received the NS intervention in the Spring will be recruited to participate in the participant interviews based on their quantitative assessment scores. The research team will recruit participants who are interested in being interviewed. Each participant will complete an individual, 30-60-minute interview intended to identify personal impacts of participation in the NS program on self-esteem, resilience, cultural identity, and substance use. Interview questions are included in an attachment Who: Interviews will be conducted by the research assistants who have received training in interview procedures.

Where: Interviews will be held in private rooms at the research site - the SRPMIC Way of Life Facility How/What data: Interview data will be collected with a digital recorder. How Long: Each interview will last for 30-45 minutes Duration: Spring interviews will be completed between May-June 2025

Step 6: Fall 2025 Usual Programming

6.1 Both groups (SRPMIC and PYT) will receive control or "usual" programming. Usual programming includes a life skills program that focuses on financial wellness for teens, called "Money Matters" (Usual Practice). Participants will learn valuable financial life skills.

Who: Control sessions will be facilitated by the research site partner (after-school program employees) who typically implement their usual programming Where: Control sessions will be held at the research site - the SRPMIC Way of Life Facility and the PYT Boys & Girls Clubs How Long: Each control session will last for 60-90 minutes, once a week for 10 weeks Duration: The Fall Usual Programming will take place from August 2025 - December 2025

Step 7: Follow-Up Assessment - Time 2 (T2) and Time 3 (T3)

7.1 SRPMIC participants will take the T3 assessment in December 2025 and PYT participants will take the T2 assessment also in Drcember 2025. Surveys will be conducted virtually on participant cell phones. The research team will also print out multiple hard copies of the survey for participants who do not have access to a cell phone. Participants will sit at individual desks that are spaced so they cannot see each other's assessment answers to minimize confidentiality risks.

Who: Virtual surveys will be administered by the PI and research team. Where: T3 and T2 assessments will be completed at the research sites - the SRPMIC Way of Life Facility and the PYT Boys & Girls Club How Long: T2 and T3 assessments will take 20-30 minutes to complete. How/What data: T2 and T3 assessment data will be collected virtually through REDCap.

Duration: The T2 and T3 assessments will be completed in December 2025

Step 8: Spring 2026 Intervention

8.1 The wait-list group (PYT) will receive the intervention (NS program). Each intervention session is based on an Indigenous cultural value and cultural activity/practice that is specific to the PYT. The PYT intervention curriculum will be developed between March 2025-December 2025. It will have a similar organizational structure.

Who: Intervention sessions will be facilitated by local cultural knowledge holders. At least one member of the research team will attend each session to ensure fidelity Where: Intervention sessions will be held at the research site - PYT Boys & Girls Club How Long: Each intervention session will last for 60-90 minutes, once a week for 10 weeks Duration: The Spring 2026 intervention will take place from January-May 2026.

8.2 The research team will take candid pictures during the intervention that can be used for results dissemination. Any identifiable pictures with youth who do not have signed assent/consent forms will be immediately deleted.

Step 9: Follow-Up Assessment - Time 3 (T3)

9.1 PYT participants will take the T3 assessment in May 2026. Surveys will be conducted virtually on participant cell phones. The research team will also print out multiple hard copies of the survey for participants who do not have access to a cell phone. Participants will sit at individual desks that are spaced so they cannot see each other's assessment answers to minimize confidentiality risks.

Who: Virtual surveys will be administered by the PI and research team. Where: T3 assessment will be completed at the research site - the PYT Boys & Girls Club How Long: T3 assessment will take 20-30 minutes to complete. How/What data: T3 assessment data will be collected virtually through Qualtrics.

Duration: T3 assessment will be completed in May 2026.

Step 10: Participant interviews

10.1 PYT Participants who received the NS intervention in Spring 2026 will be recruited to participate in the participant interviews based on their quantitative assessment scores. The research team will recruit participants who are interested in being interviewed. Each participant will complete an individual, 30-60-minute interview intended to identify personal impacts of participation in the NS program on self-esteem, resilience, cultural identity, and substance use.

Who: Interviews will be conducted by the research assistants who have received training in interview procedures.

Where: Interviews will be held in private rooms at the research site - the PYT Boys & Girls Club How/What data: Interview data will be collected with a digital recorder. How Long: Each interview will last for 30-45 minutes Duration: Fall interviews will be completed between May-June 2026

ELIGIBILITY:
Inclusion:

* English-speaking
* Currently in grade 7-12 at time of enrollment
* Member of the Salt River Pima Maricopa Indian Community (SRPMIC) OR member of the Pascua Yaqui Tribe (PYT)
* Engaged in after school programs.

Exclusion:

• Non-American Indians will be excluded from statistical analysis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Past 30-Day Substance Use | Baseline, Immediately Post-Invervention, 3 months follow-up post-intervention
  Data collection will focus on recent, self-reproted (past 30-day) use frequency of alcohol, cigarettes/e- cigarettes, marijuana, and other hard drugs (crystal methamphetamine, cocaine, etc.). The survey will also include a qualifying question on lifetime use of the following substances in order to measure delay of onset of use (in the case that participants have never used any of the measured substances).
Rosenberg Self-Esteem Scale | Baseline, Immediately Post-Invervention, 3 months follow-up post-intervention
  Self-Reported measure of self-esteem using the Rosenberg self-esteem scale. The is scored by totaling the individual 4-point items after reverse-scoring the negatively worded items with a minimum score of 10 and maximum score of 40. Higher scores indicate a better outcome (stronger sense of self-esteem).
Child and Youth Resilience Measure | Baseline, Immediately Post-Invervention, 3 months follow-up post-intervention
  Self-Reported measure of resilience using the Child and Youth Resilience Measure. The items within the measures can be directly summed to gain a total score of an individual's resilience. Responses are on a 5-point Likert scale (going from 1-5), the minimum score is 17 and the maximum score is 85. Higher scores indicate a better outcome (stronger sense of resilience).
Cultural Efficacy | Baseline, Immediately Post-Invervention, 3 months follow-up post-intervention
  Self-Reported measure of cultural efficacy. This is on a 5-point Likert scale with a minimum score of 8 and maximum score of 40. Higher scores indicate a better outcome (cultural efficacy).
Awareness of Connectedness Scale | Baseline, Immediately Post-Invervention, 3 months follow-up post-intervention
  Self-Reported measure of awareness of connectedness to culture using the Awareness of Connectedness Scale. This is a 3-point Likert scale with scores ranging from 12 to 36. Higher scores indicate a better outcome (stronger awareness of connectedness).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Hunter, PhD, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - Way of Life Facility, Scottsdale, Arizona
  - Pascua Yaqui Tribe Boys & Girls Club, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No
This study includes data collection with two sovereign Native Nations in Arizona. Collected data and access to this data is ultimately under the discretion of the Tribal leadership, the departments involved, and the Office of the Attorney General.